CLINICAL TRIAL: NCT07232160
Title: Is DSA Display Along With Bispectral Index Superior to the Display of Bispectral Index Alone in Detecting Emergence From Propofol and Opiate Anesthesia? A Prospective Observational Study in Patients Older Than 65 Years?
Brief Title: Is Density Spectral Array Display Along With Bispectral Index Superior to the Display of Bispectral Index Alone
Acronym: DSA-Light
Status: Not yet recruiting | Type: Observational
Sponsor: The University of Queensland (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 2025/HE000173
Record Dates: First submitted 2025-08-29; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-08

CONDITIONS: Awareness During General Anesthesia
Keywords: depth of anaesthesia monitoring; processed EEG; EEG; density spectral array; Bispectral index; older adults; patients older than 65 years; general anaesthesia; total intravenous anaesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Primary cohort: * Age ≥ 65 years undergoing elective procedures of 1-3 hours' duration requiring GA.
  * Procedures in which a DoA monitor can be applied to the forehead.
  * Patients receiving intravenous propofol and opiate anesthesia using supraglottic airway device.
  * Patient able to provide informed consent.
  Interventions: Device: Depth of anesthesia monitoring using processed EEG

INTERVENTIONS:
Device: Depth of anesthesia monitoring using processed EEG — Comparison of processed EEG monitor (Bispectral index) with and without Density spectral array

SUMMARY:
A study to evaluate the use of density spectral array display in comparison with Bispectral index in a clinical setting.

DETAILED DESCRIPTION:
Propofol-based total intravenous anesthesia (TIVA) is a popular general anesthesia (GA) technique with an increased risk of unintended awareness under GA, which can be a devastating and life-changing complication. Age-related changes may impact the performance of EEG-derived depth of anesthesia indices in those older than 65 years, particularly in the presence of cognitive disorders.

Hypothesis: In comparison to monitor 1 (BIS only), monitor 2 (DSA + BIS) will have higher sensitivity and specificity to detect recovery

Objectives:

Investigators will prospectively measure the sensitivity and specificity of monitor 1 versus monitor 2 in patients older than 65 years receiving propofol-based TIVA.

Methods:

Investigators will recruit 70 participants from the Royal Brisbane and Women's Hospital (RBWH) who are aged 65 years or older and scheduled for elective endovascular or endoscopic urologic procedures.

Investigators aim to determine whether the display of DSA can enhance the sensitivity and specificity of depth of anesthesia monitors in detecting sudden changes in anesthetic depth in older patients. This may enhance the detection of inadequate administration or delivery of propofol and may lower the incidence of unintended awareness under general anesthesia in that age group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years undergoing elective procedures of 1-3 hours' duration requiring GA.
* Procedures in which a DoA monitor can be applied to the forehead.
* Patients receiving intravenous propofol and opiate anaesthesia using supraglottic airway device.
* Patient able to provide informed consent.

Exclusion criteria:

* Administration of ketamine/dexmedetomidine.
* Administration of inhaled anaesthetic agents or nitrous oxide
* Administration of muscle relaxation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: • Age ≥ 65 years undergoing elective procedures of 1-3 hours' duration requiring GA at RBWH
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
aim | In the perioperative period, following the cessation of anesthesia, the patient begins to emerge from a deep anesthetic state to a lighter state and then regains consciousness. The time frame is usually in minutes, but varies depending on various factors
  Sensitivity and specificity of Bispectral index combined with density spectral array compared with Bispectral index alone in detection of emergence from general anesthesia. Emergence from anaesthesia manifests in changes in the BIS and/or DSA suggestive of a change in the depth of anesthesia and progress towards regaining consciousness.
Primary aim | In the perioperative period, time following the cessation of intravenous anesthesia after the procedure; emergence from anesthesia usually takes place over a few minutes to hours.
  Evaluate the sensitivity and specificity of Bispectral index combined with density spectral array compared with Bispectral index alone in the detection of the timing of emergence from general anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boules, MB BCh, Principal Investigator — The University of Queensland
Locations (1):
- Royal Brisbane and Women's Hospital, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided
The data collected is owned by Metro North Health and I need their approval before doing so